CLINICAL TRIAL: NCT02784548
Title: Adapting Virtual Reality Technology for the Treatment of Phantom Limb Pain
Brief Title: Virtual Reality for Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1729-P
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality (Experimental): Using a Virtual reality (VR) headset, motion sensors, and VR software, the investigators will create a customized VR treatment for each participant that engages them in movements and exercises involving their missing limb in a game-like environment. For example, participants may use the headset to engage in activities such as driving a race car around a course requiring both arms, ski down simulated slopes, or manipulate objects.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Using a VR headset, motion sensors, and VR software, the investigators will create a customized VR treatment for each participant that engages them in movements and exercises involving their missing limb in a game-like environment. For example, participants may use the headset to engage in activities such as driving a race car around a course requiring both arms, ski down simulated slopes, or manipulate objects.

SUMMARY:
This study will develop a virtual reality-based treatment for phantom limb pain among Veterans and test it against the most established behavioral therapy for phantom limb pain, mirror therapy.

DETAILED DESCRIPTION:
The VA system performs more than 10% of all amputations in the U.S., a percentage translating into more than 50,000 upper and lower extremity amputations in the past decade. Among Veterans with amputations, research suggests that upwards of 70% experience phantom limb pain (PLP), an often chronic and debilitating condition with adverse effects on quality of life and poor responsiveness to conventional pain treatments. The use of virtual reality technology for chronic pain management is a novel and rapidly advancing area of study, with existing research suggesting that virtual reality treatments are effective for acute pain management, promising for chronic pain management, and as yet untested for PLP. In the current study, the investigators will develop a virtual reality environment that simulates mirror therapy - the gold standard behavioral treatment for PLP - comparing the efficacy of this modality in a population of Veterans with PLP against a standard mirror therapy treatment validated by this research team in a previously supported clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-75 Veteran receiving care at VA San Diego Healthcare System
* Upper or lower extremity amputation with reported PLP for at least six months
* PLP intensity > 3/10
* English-speaking, literate, with stable residence
* Able to operate a VR headset as evidenced by direct observation

Exclusion Criteria:

* Major medical illness that might confound effects of pain on function, e.g.:

  * advanced cardiac
  * pulmonary disease
* current active alcohol or substance use disorder as evidenced from medical record
* currently active suicidality
* homicidality, or unstable psychiatric status in previous three months as measured by direct observation, patient self-report, or medical record
* moderate or severe cognitive impairment as demonstrated by medical diagnosis or clinical observation
* prior mirror therapy experience

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Rutledge, PhD MA, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Phantom Limb Pain Questionnaire (PLPQ)
Description: The PLPQ assesses the severity of PLP, stump pain and phantom limb sensation. Severity is assessed on a standard 11-point Likert scale pain measure, range 0-10 with higher scores indicating greater PLP.
Time Frame: PLPQ scores before versus after initial use of the VR treatment in the laboratory
Population: Veterans with PLP. The mirror therapy group was a pre-specified control group that was not completed due to recruitment challenges.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mirror Therapy: Mirror Therapy comparison group
Arm/Group | Virtual Reality | Mirror Therapy
Number analyzed (Participants) | 15 | 0
units on a scale
  Pre-VR use | 1.2 (1.6) |
  Post-VR use | .5 (.94) |

ADVERSE EVENTS:
Time Frame: During participation, up to 1 year
Arm/Group | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
As noted in the results section, this study did not contain long-term follow-up or enroll the a prior planned mirror therapy control group due to recruitment limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02784548/Prot_SAP_000.pdf